CLINICAL TRIAL: NCT04807257
Title: A First-in-Human Study of Auger Molecular Therapy (AMT) in Patients With Malignant Cutaneous Lesions From Advanced Solid Tumors
Brief Title: Auger Molecular Therapy (AMT) for Malignant Cutaneous Lesions Treatment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NanoRay Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT-NR-33
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Malignant Fungating Wound
Keywords: Malignant fungating wound; Malignant wound; Malignant cutaneous lesion

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Malignant Cutaneous Lesions from Advanced Solid Tumors (Experimental): The IUdR, which is manufactured as lyophilized powder for injection, is dissolved by normal saline before use.
  There are three cohorts with escalating doses of IUdR starting from an injection dose of 0.1 mL per lesion surface area unit of 1 cm2 and if tolerated, escalate to 0.2 mL/cm2 and to 0.25 mL/cm2 as presented below. Meanwhile, the upper limit of total injection doses of IUdR in the 3 levels are 2.83, 5.65, and 7.07ml , which correspond to 0.059, 0.118, and 0.147 mg/kg for a 60 kg adult, respectively. The dose of AUTRON Therapy System irradiation for all 3 cohorts keeps fixed at 25 Gy over 5 days (5 Gy/day).
  Interventions: Combination Product: Auger Molecular Therapy (AMT)

INTERVENTIONS:
Combination Product: Auger Molecular Therapy (AMT) — The AMT consists of intratumorally delivered IUdR and local irradiation via AUTRON Therapy System.

SUMMARY:
This is a first-in-human, single-arm, open-label, dose escalating study to determine the safety and the recommended maximum tolerated dose of the AMT in subjects with malignant cutaneous lesions.

AMT is a combination therapy of a drug (IUdR) and a device (AUTRON Therapy System). IUdR is an iodinated thymidine analogue that is preferentially incorporated into DNA in rapid growing cells. The AUTRON Therapy System generates characteristic X-Ray photons around 33.4 keV, matching the K-edge energy of Iodine (33.17 keV), which can efficiently induce Auger electron emissions from IUdR in cancer DNA, resulting in extensive DNA damage and cancer cell death.

DETAILED DESCRIPTION:
NanoRay Biotech is developing a novel investigational therapeutic system called Auger Molecular Therapy (AMT), which consists of a drug, Iododeoxyuridine (IUdR), and a medical device, AUTRON Therapy System, intended for the palliative treatment of malignant cutaneous lesions. IUdR is an iodinated analogue of deoxyuridine, which can be incorporated into DNA of cancer cells because it is a thymidine analogue. The AUTRON Therapy System is a complete, standalone low energy X-Ray radiation source (80 kVp, 100 μA) intended for local irradiation. The AUTRON Therapy System contains a novel design of transmission type X-Ray tube, which allows electron beams to pass through the metal target and generates characteristic X-Ray similar to synchrotron radiation.

The combination product is intended to induce Auger effect to augment the damage on tumor cells, while lowering the adverse effect on normal cells. IUdR is an iodinated thymidine analogue that is preferentially incorporated into DNA in rapid growing cells (such as cancer cells) after administration. The AUTRON Therapy System generates characteristic X-Ray photons around 33.4 keV, matching the K-edge energy of Iodine (33.17 keV), which can efficiently induce emissions of Auger electrons when hitting the Iodine atoms on IUdR in cancer DNA, resulting in extensive DNA damage and cancer cell death. Furthermore, the characteristic X-Ray photons generated by the AUTRON Therapy System have a low penetration rate in biological materials, which give the maximum dose on superficial lesions and much reduced dose on peripheral or deep normal tissues, fitting the need on the management of malignant cutaneous lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Histologically confirmed diagnosis of advanced head and neck cancers, breast cancers, gastrointestinal cancers, pancreatic cancers, gallbladder cancer, liver cancers, endometrial cancer, and/or prostate cancers.
3. Cutaneous lesion(s) that is (are) from distant metastasis or direct invasion of tumor types as above.
4. The size of lesion to be treated can be covered by the irradiation Applicator (a circle in the diameter of 6 cm, around 28.27 cm2 in surface area).
5. The subject must have malignant cutaneous lesion thickness of ≤0.7 cm
6. The subject must have measurable disease by the square grid methods using transparency wound dressing or projection light.
7. ECOG Performance Status ≤ 3.
8. Adequate organ functions determined within 4 weeks prior to enrollment defined as:

   * Hematologic: (ANC) ≥ 1.0 × 109/L; Hemoglobin ≥ 9 g/dL; Platelet count ≥ 100 × 109/L; PT or PTT ≤ 1.5 ×upper limit of normal value (ULN).
   * Hepatic function: bilirubin < 2 × ULN, and AST and ALT < 3 × ULN.
   * Renal Function: creatinine clearance > 50 mL/min.
9. Provided written informed consent in accordance with all applicable regulations and followed the study procedures.
10. Subjects are capable of understanding the investigational nature, potential risks and benefits of the study.
11. A subject who is receiving concurrent systemic therapy, including chemotherapy and immunotherapy, can be recruited without ceasing the systemic therapy. However, the subject should be discontinued from the trial if the subject requires treatment with a new systemic therapy.

Exclusion Criteria:

1. Restless patients who are unable to lie or sit in a cast for 25 mins.
2. Hypersensitive to the study drug.
3. Patients with connective tissue diseases
4. Patients with known syndromes associated with radiation sensitivity.
5. Patients with prior radiotherapy to the area which could compromise safety of additional treatments.
6. Lesion(s) that is derived from localized and curable tumor(s).
7. Lesion(s) with friable surface or necrotic changes.
8. Lesion(s) locates on the eyelid, the eye, the genitalia, the lip and near the carotid artery that might expose the patients in a great risk when receiving irradiation.
9. Uncontrolled intercurrent illness, such as severe infection, symptomatic heart disease, etc.
10. Concomitant treatment with therapeutic anticoagulants.
11. Receiving or requiring immunosuppressive therapies.
12. Human immunodeficiency virus (HIV) infection.
13. Any underlying medical conditions, which in the opinion of the investigator, would make the study hazardous or make it difficult to monitor adverse effects.
14. Participation in any investigational drug study within 4 weeks prior to screening.
15. Pregnant or breast-feeding female. Note: Confirmation that women of child- bearing potential are not pregnant. A negative serum or urine β-human chorionic gonadotropin (β-hCG) pregnancy test result is to be obtained during the screening period.
16. Fertile males and females who are unwilling to employ adequate means of contraception (e.g., condom with spermicide, diaphragm with spermicide, birth control pills, injections, patches, or intrauterine device) during the study and through 4 to 6 months after the study.
17. Patients with a QTcF >470 ms on screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lesion severity | 56 weeks from Day -1 predose
  In this trial, local lesion assessment will be carried out by a simplified Modified Severity Weighted Assessment Tool (mSWAT) without %BSA parameter, since the AMT is applied only on local and single lesion. A local skin scoring by area with a multiplication by weighting factors of various lesion types (patch=1, plaque=2 and tumor=4) is applied for mSWAT evaluation.
Improvement of quality of life | 8 weeks from Day -1 predose
  The Taiwanese version of the McGill Quality of Life Questionnaire (MQOL) consists of 16 items, global QOL questions and open-ended questions allowing patients to self-report life events that have influenced their QOL. There are four parts in MQOL: physical symptoms (items 1-4), psychological well-being (items 5-8), existential well-being (items 9-14), and support issues (items 15 and 16). All of the response categories are based on a numerical scale of from 0 to 10. The all score will be divided into four parts and a high score indicates a better QOL.
Assess the drug safety during treatment | 4 weeks of treatment cycle
  Safety evaluation will be based on the percentage of subjects with dose-limiting toxicity (DLT), adverse events (AE), and serious adverse events (SAE). Toxicity will be classified by National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Assess the drug safety post-treatment | 4 weeks post treatment
  Safety evaluation will be based on the percentage of subjects with dose-limiting toxicity (DLT), adverse events (AE), and serious adverse events (SAE). Toxicity will be classified by National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Local control of lesion | 12 weeks
  The lesion condition change is evaluated by CT before and after treatment.

SECONDARY OUTCOMES:
Systemic immune response | 56 weeks
  Evaluated by changes in composition of peripheral lymphocytes in patient blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

REFERENCES:
- See also: The principal of Auger Molecular Therapy — https://nanoray.com/e/%e5%88%86%e5%ad%90%e6%b2%bb%e7%99%82-%e5%8e%9f%e7%90%86e/